CLINICAL TRIAL: NCT05209568
Title: Changes in Serum IL-2 Levels Following a Single Oral Dose of Gluten
Brief Title: Immune Responses to Gluten
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Children's Hospital Colorado (Other); Celiac Disease Foundation (Unknown)
Responsible Party: Principal Investigator, Jocelyn Silvester, Director of Research, Celiac Disease Program, Boston Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P00039708
Record Dates: First submitted 2022-01-13; First posted 2022-01-26 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Celiac Disease; Malabsorption Syndromes; Digestive System Disease; Intestinal Disease; Gastrointestinal Diseases; Gluten Sensitivity; Celiac Disease in Children
Keywords: gluten; cytokine; T cell immune response
MeSH Terms: conditions — Celiac Disease; Malabsorption Syndromes; Digestive System Diseases; Intestinal Diseases; Gastrointestinal Diseases

STUDY DESIGN:
Intervention Model Description: This is a multi-center study of immune responses to gluten in persons with celiac disease and healthy controls. All participants will have baseline blood drawn to assess immune responses at baseline in addition to four hours after a single oral dose of gluten.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Celiac Disease (Experimental): Individuals with a confirmed diagnosis of celiac disease based on serology and/or histology
  Interventions: Dietary Supplement: Gluten Powder
- Healthy Controls (Experimental): Individuals without a diagnosis of celiac disease
  Interventions: Dietary Supplement: Gluten Powder

INTERVENTIONS:
Dietary Supplement: Gluten Powder — Single oral dose of gluten powder

SUMMARY:
This is a study of immune responses after eating gluten powder in people with celiac disease and healthy controls.

DETAILED DESCRIPTION:
This is a multi-site open-label single dose gluten challenge study. Participants will provide a blood sample for measurement of cytokines before and 4 hours after eating gluten powder.

ELIGIBILITY:
Inclusion Criteria:

1. On a gluten-free diet for ≥ 4 weeks
2. Willing to consume gluten for research
3. For the celiac disease arm, diagnosis confirmed by serology and/or histology

Exclusion Criteria:

1. Pregnancy
2. Wheat allergy
3. Type 1 diabetes
4. BMI z-score < -2
5. History of more than minimal symptoms following gluten exposure on a gluten-free diet
6. Comorbid condition that in the opinion of the investigator would interfere with study participation or would confound study results

Ages: 2 Years to 101 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in serum interleukin-2 (IL-2) level from baseline to 4 hours after a single oral dose of gluten | Baseline, 4 hours
  To determine the change in serum IL-2 level from baseline after a single oral dose of gluten

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn A Silvester, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (2):
- United States (2):
  - Children's Hospital Colorado, Aurora, Colorado
  - Boston Children's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Individual participant demographic and cytokine data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal

REFERENCES:
- [Background] Goel G, Tye-Din JA, Qiao SW, Russell AK, Mayassi T, Ciszewski C, Sarna VK, Wang S, Goldstein KE, Dzuris JL, Williams LJ, Xavier RJ, Lundin KEA, Jabri B, Sollid LM, Anderson RP. Cytokine release and gastrointestinal symptoms after gluten challenge in celiac disease. Sci Adv. 2019 Aug 7;5(8):eaaw7756. doi: 10.1126/sciadv.aaw7756. eCollection 2019 Aug. PMID 31457091
- [Background] Goel G, Daveson AJM, Hooi CE, Tye-Din JA, Wang S, Szymczak E, Williams LJ, Dzuris JL, Neff KM, Truitt KE, Anderson RP. Serum cytokines elevated during gluten-mediated cytokine release in coeliac disease. Clin Exp Immunol. 2020 Jan;199(1):68-78. doi: 10.1111/cei.13369. Epub 2019 Oct 1. PMID 31505020
- [Background] Tye-Din JA, Daveson AJM, Ee HC, Goel G, MacDougall J, Acaster S, Goldstein KE, Dzuris JL, Neff KM, Truitt KE, Anderson RP. Elevated serum interleukin-2 after gluten correlates with symptoms and is a potential diagnostic biomarker for coeliac disease. Aliment Pharmacol Ther. 2019 Oct;50(8):901-910. doi: 10.1111/apt.15477. Epub 2019 Sep 4. PMID 31483515